CLINICAL TRIAL: NCT04824807
Title: The Comparison of the Effects of Clinical Pilates and Yoga Training in Women With Lymphedema After Breast Cancer
Brief Title: Effects of Clinical Pilates and Yoga Training in Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ferdiye Zabit, MSc physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-2020-0103
Record Dates: First submitted 2021-03-10; First posted 2021-04-01 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Lymphedema; Exercise
Keywords: Pilates; Yoga; Volumetric measurement; Muscle Strength Dynamometer; Respiratory Function Tests
MeSH Terms: conditions — Lymphedema; Motor Activity | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical Pilates Group (Experimental): Individuals in the this group will receive 24 sessions of Clinical Pilates training 3 times a week for 8 weeks. During the training, individuals will be asked to wear compression stockings during the 8 weeks. An educational booklet will be given to the each group.
  Interventions: Other: Clinical Pilates; Other: An educational booklet
- Yoga Group (Experimental): Individuals in the this group will be given 24 hours of yoga training 3 times a week for 8 weeks. During the training, individuals will be asked to wear compression stockings during the 8 weeks. An educational booklet will be given to the each group.
  Interventions: Other: Yoga; Other: An educational booklet
- Control Group (Other): Individuals in the this group will not receive any treatment. Individuals will be asked to wear compression stockings during the 8 weeks. An educational booklet will be given to the each group.
  Interventions: Other: An educational booklet

INTERVENTIONS:
Other: Yoga — The yoga classes included a progression of low-impact, modified poses, stretching and isometric exercises focused on the shoulders, arms, and chest, and meditation. Breathing and poses to drain the lymphatic system were incorporated throughout the yoga practice to assist with lymphatic flow.
  Exercises: sitting down badrasana, ardha navasana, dhanurasan, setu bandhasana, Urdhva Dhanurasana, Urdhvamukha Svanasana, Virabhadrasana, Warrior Virasana, Supta Virasana, Surya Namaskar, Mayurasana, Padmasana, Bharadvajasana.
  Other Names: Exercises program
  Arms: Yoga Group
Other: Clinical Pilates — before starting the clinical Pilates exercise program, the patients were trained on Pilates exercises and postures. During training, the patients were taught how to create lumbopelvic stability (core stabilization), which is the basis for Pilates exercises, and spinal stabilization and appropriate posture techniques.
  Exercises: cork screw, toy soldier, kleopatra, the saw,breast stroke preparation, swimming, diamond press - arm openings, scapula isolations, open book, scissors, shoulder bridge.
  Other Names: Exercises program
  Arms: Clinical Pilates Group
Other: An educational booklet — Only educational booklets will be given to the control group
  Other Names: No treatment

SUMMARY:
The aim of our study is to compare the effects of clinical Pilates and yoga training on lymphedema, upper limb muscle strength, proprioception, functions and quality of life in women with lymphedema after breast cancer.

DETAILED DESCRIPTION:
A total of 60 post breast cancer lymphedema individuals will be included in our study. The study will be performed in individuals who live in T.R.N.C and who develop mild, moderate or severe lymphedema after breast cancer in the 35-70 age range.

A randomized controlled trial design with three groups were used; 1) A Hatha yoga intervention group, 2) Clinical Pilates intervention group, 3) Control group.

Individuals in the intervention groups will be given 24 sessions of yoga or Clinical Pilates training 3 times a week for 8 weeks. Control group will not receive any treatment. During the training, and control group individuals will be asked to wear compression stockings during the 8 weeks and an educational booklet will be given to the each group.

The yoga classes included a progression of low-impact, modified poses, stretching and isometric exercises focused on the shoulders, arms, and chest, and meditation. Breathing and poses to drain the lymphatic system were incorporated throughout the yoga practice to assist with lymphatic flow. Before starting the Clinical Pilates exercise program, the patients will be trained on Pilates exercises and postures. During training, the patients will be taught how to create lumbopelvic stability (core stabilization), which is the basis for Pilates exercises, and spinal stabilization and appropriate posture techniques.

As a result of the research, the data will be analyzed to determine which treatment method is more effective in lymphedematous individuals.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors,
* who are between the ages of 35-70,
* who have unilateral mild, moderate or severe
* lymphedema in the upper extremities after breast cancer treatment,
* who have taken any of the Lymphedema treatment methods at least 6 months ago will be included.

Exclusion Criteria:

* Presence of metastatic breast cancer,
* Currently receiving adjuvant therapy (chemotherapy, radiotherapy, hormone therapy),
* Severe heart failure (Class III),
* Infections in extremities (fungal, redness, temperature increase),
* Severe pain in the axillary region (eg: axillary web syndrome,
* reflex sympathetic dystrophy, neuropathy),
* Persons participating in a regular exercise program in the last 6 months will be excluded from the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
upper extremity lymphedema | eight weeks
  Bilateral arm volume was measured with the upper extremity volumetric cup.Participants submerged their arm and hand into a water-filled column up to their axilla, and the volume of displaced water was recorded. Due to differences in volumetric measurement between both arms, it will be recorded.

SECONDARY OUTCOMES:
upper extremity muscle endurance | eight weeks
  Muscle endurance will be evaluated by isokinetic dynamometer.For the extremity to be tested in the supine position, when the shoulder is in 90° abduction and the elbow is 90° flexed, the isokinetic force measurements of the shoulder internal and external rotation movements will be performed with an angular velocity of 240° / s at 15 repetitions.
upper extremity muscle strength | eight weeks
  muscle strength will be evaluated by isokinetic dynamometer.For the extremity to be tested in the supine position, when the shoulder is in 90° abduction and the elbow is 90° flexed, the isokinetic force measurements of the shoulder internal and external rotation movements will be performed with an angular velocity of 180° / s at 5 repetitions.
upper extremity proprioception | eight weeks
  upper extremity proprioceptionuwill be evaluated by isokinetic dynamometer. Proprioception tests were performed during active joint position sense, passive joint position sense and kinesthesia.
  While the individuals are lying on their back, the shoulder will be positioned in 90° abduction in the coronal plane and the elbow in 90° flexion and fixed at the level of the chest and ankle. proprioception test, subjects were testedwhile lay comfortably down an adjustable bed. To eliminate visual clues and ears closed with headphones to all subjects were blindfolded.shoulder active joint position sense, passive joint position sense and kinesthesia test measurements of 0-45° external rotation movements will be performed with the shoulder in of 90° abduction and the elbow 90° in flexion positıon, with to be 3 repetitions. A pressure splint will be worn to prevent sensory input to the skin in passive joint position sense.
upper extremity functions | eight weeks
  to evaluate upper extremity functions will be done DASH questionnaire.This survey is a disability and symptom scale that evaluates the upper extremity functions in the last week. It contains 30 items regarding symptoms and daily life activities. 21 items provide information about levels of difficulties experienced with the shoulder, arm and hand while carrying out different physical activities, 5 items provide information about pain, tingling, weakness and stiffness during physical activities of differing intensity, and 4 items provide information about social activities, occupation and sleeping disorders. DASH survey scores an a 5-point likert scale and total scores changes in the range of 0-100. It is completed in about 5-7 minutes. The score. A higher score indicates more disabilities and symptoms.
Quality of Life Questionnaire | eight weeks
  to evaluate Quality of Life Questionnaire will be done EORTC QLQ-BR23. It is a 4-point Likert scale ranging from 1 (not at all) to 4 (very much). The total high scores obtained from the QLQ-BR 23 questionnaire with which patients' quality of daily lives is analyzed indicate difficulties in performing daily living activities, functional activities and reduction in the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus